CLINICAL TRIAL: NCT04441060
Title: Development of a Suicide Risk Scale and Distress Intervention for the Patients With Chronic Medical Illness or Physical Disabilities
Brief Title: Suicide Risk Scale and Distress Intervention for the Patients With Chronic Medical Illness or Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pusan National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL19C0039
Record Dates: First submitted 2020-04-23; First posted 2020-06-22 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2022-05

CONDITIONS: Chronic Illnesses; Physical Disability
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- distress intervention subject group (Experimental): Distress intervention program will be developed, and applied to the subject group, and they will be assessed before and after the intervention program with several tools.
  Interventions: Other: Distress intervention (CBT & Mindfulness-based program)
- distress intervention control group (No Intervention): No intervention will be applied to the control group. They will be assessed before and after the intervention program with same tools with subject group.

INTERVENTIONS:
Other: Distress intervention (CBT & Mindfulness-based program) — Distress intervention is not fully developed yet, but we are working on the development of distress intervention based on CBT & Mindfulness-based program.
  Arms: distress intervention subject group

SUMMARY:
The aims of this study are developments of distress intervention and a suicidal risk scale for the patients with chronic medical illness or physical disabilities. To do these things, four times of interview & completion of self-report scale will be done, and newly developed distress intervention will be simulated to subject group and control group.

DETAILED DESCRIPTION:
The aims of this study are developments of distress intervention and a suicidal risk scale for the patients with chronic medical illness or physical disabilities.

To achieve the aims, multidisciplinary team is organized such as doctors of internal medicine, rehabilitative medicine, psychiatrist specialized in psychosomatics, psychologist, nurse, social worker and researchers.

Before developing the intervention and scale, review of literature about intervention, suicide, management system of chronic illness, several scales and others are done. Also, qualitative interview and self report scale with those patients are done to figure out what bothers them most, how they feel, and what kind of help they need.

Based on collected data, means of intervention is carefully selected and further review of literature is proceeded. Also, questions which describe patients' feeling, discomfort, and need are made. Moreover, modified management system of chronic illness is planned to develop to link between those who need help among patients and multidisciplinary team members.

Once, the intervention is developed, subject group and control group are recruited in stroke patients, and the intervention is simulated. The change of distress is measured before and after the intervention, and 1 month later the intervention is finished with several tools such as WHOQOL-BREF, Perceived Stress Scale, Rosenberg Self-Esteem Scale, Acceptance of Disability Scale, Participation Scale, Pain Belief & Perception Inventory, Insomnia Severity Index, FACIT-Fatigue, Hospital Anxiety and Depression Scale, digit span, trail making test, stroop test, verbal fluency test.

Also, newly developed questions and other scales are performed among patients to determine whether the newly developed questions are appropriate and how well they reflect their difficulties and feelings. After selecting the appropriate questions, the revised version will be tested by the patients twice in a different time frame.

If the revised version is appraised appropriate, it will be distributed as a cell phone application.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic illness or physical disabilities (Heart failure, Chronic kidney disease, Stroke patients)

Exclusion Criteria:

* Patients who have other severe illness such as cancer, severe memory impairment or intellectual disabilities and others

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Quality of life: World Health Organization's quality of life instrument -short version (WHOQOL-BREF) | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Quality of life was assessed three times using the World Health Organization's quality of life instrument - short version (WHOQOL-BREF); before and after the intervention, and 1 month later after the intervention is finished. The amount of quality of life change will be one of the primary outcomes.
Stress: Perceived Stress Scale (PSS-10) | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Stress was assessed three times using Perceived Stress Scale (PSS-10); before and after the intervention, and 1 month later after the intervention is finished. The amount of Stress change will be one of the primary outcomes.
Resilience: Connor-Davidson Resilience Scale (CDRS) | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Resilience was assessed three times using Connor-Davidson Resilience Scale (CDRS); before and after the intervention, and 1 month later after the intervention is finished. The amount of resilience change will be one of the primary outcomes.
Self-esteem: Rosenberg Self-Esteem Scale | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Self-esteem was assessed three times using Rosenberg Self-Esteem Scale; before and after the intervention, and 1 month later after the intervention is finished. The amount of Self-esteem change will be one of the primary outcomes.
Acceptance of disability: Acceptance of Disability Scale | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Acceptance of disability was assessed three times using Acceptance of Disability Scale; before and after the intervention, and 1 month later after the intervention is finished. The amount of acceptance of disability change will be one of the primary outcomes.
Social participation: Participation Scale | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Social participation was assessed three times using Participation Scale; before and after the intervention, and 1 month later after the intervention is finished. The amount of Social participation change will be one of the primary outcomes.
Pain: Pain belief & Perception inventory (PBPI) | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Pain was assessed three times using Pain belief & Perception inventory (PBPI); before and after the intervention, and 1 month later after the intervention is finished. The amount of pain change will be one of the primary outcomes.
Insomnia: Insomnia Severity Index (ISI) | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Insomnia was assessed three times using Insomnia Severity Index (ISI); before and after the intervention, and 1 month later after the intervention is finished. The amount of Insomnia change will be one of the primary outcomes.
Fatigue: FACIT-Fatigue | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Fatigue was assessed three times using FACIT-Fatigue; before and after the intervention, and 1 month later after the intervention is finished. The amount of fatigue change will be one of the primary outcomes.
Depression, Anxiety: Hospital Anxiety and Depression Scale | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Depression and anxiety was assessed three times using Hospital Anxiety and Depression Scale; before and after the intervention, and 1 month later after the intervention is finished. The amount of depression and anxiety change will be one of the primary outcomes. The 14-item Hospital Anxiety and Depression Scale comprises two subscales assessing anxiety and depression. Participants were asked to rate each item on a 4- point Likert scale (0-3); subscale scores ranged from 0 to 21. A cutoff score of 8 was applied to define clinical level of anxiety and depression.
Attention: Digit Span Test | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Attention was assessed three times using the Digit Span Test; before and after the intervention, and 1 month later after the intervention is finished. The Digit Span test is a neuropsychological test in most common use for measuring attention-concentration and working memory. The amount of Digit Span Test result (percentile score) change will be one of the primary outcomes.
Attention: Trail Making Test | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Attention was assessed three times using the Trail Making Test; before and after the intervention, and 1 month later after the intervention is finished. The Trail Making Test is a widely used neuropsychological measure that is known as a test of psychomotor speed, attention, sequencing, mental flexibility. The amount of Trail Making Test result (time to complete test) change will be one of the primary outcomes.
Attention: Stoop Color-Word Test | baseline, within a week after the end of the full course of intervention, and 1 month later after the intervention is finished
  Attention was assessed three times using the Stoop Color-Word Test; before and after the intervention, and 1 month later after the intervention is finished. The Stroop color word test is useful to examines the frontal lobe function of selective attention and inhibition. The amount of Stoop Color-Word Test results (Time taken to perform, number performed correctly, number of errors) change will be one of the primary outcomes.
Suicide risk : Korea-Suicide Risk Scale (the name can be changed later) | through study completion, an average of 1 year
  Suicide risk scale will be developed and compared with other known tools. The scale has no definite name yet, but it can be called as Korea-Suicide Risk Scale for now. A score will be reported on a scale, the higher score, the severe the suicidal risk. About 90 questions are developed for the scale, and out of them, meaningful questions will be selected through large-scale interview & comparison with other scales about suicide during the study. We are not sure how many questions are selected by now, so the minimum or maximum score cannot be decided so far. Though, the questions have 4 point scale from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Jin Hahm, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No